CLINICAL TRIAL: NCT05511844
Title: Phase I Multicenter, Open-Label, First-in-Human Study of ORM-5029 in Subjects With HER2-Expressing Advanced Solid Tumors
Brief Title: Study of ORM-5029 in Subjects With HER2-Expressing Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Orum Therapeutics USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORM-5029-01-001
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; HER-2 Protein Overexpression; HER-2 Gene Amplification; HER2 Gene Mutation
Keywords: HER2 Expressing; HER2 Positive; HER2 Associated; Antibody Drug Conjugate; Protein-Degradation; GSPT1; Celmod; Imid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): All participants receive ORM-5029 in escalating dose cohorts in Part 1 Dose Escalation and at the Expansion Dose Level (EDL) in Part 2 Dose Expansion.
  Interventions: Drug: ORM-5029
- Part 2 Dose Expansion (Experimental): All participants receive ORM-5029 at dose levels with pharmacodynamic activity or efficacy signals (Expansion Cohort A) or at the Expansion Dose Level (EDL) (Expansion Cohorts B and C).
  Interventions: Drug: ORM-5029

INTERVENTIONS:
Drug: ORM-5029 — Intravenous infusion

SUMMARY:
This is a Phase 1 first-in-human study of ORM-5029 in participants with HER2-expressing advanced solid tumors. The study consists of two parts: a Part 1 Dose Escalation and Part 2 Dose Expansion.

ELIGIBILITY:
KEY INCLUSION CRITERIA

* Have histologically confirmed advanced breast cancer that is HER2+ by In Situ Hybridization (ISH) and/or at least 1+ staining by Immunohistochemistry (IHC), determined at the institution.
* Participant is not a candidate for or would be unlikely to tolerate or derive significant clinical benefit from, appropriate standard-of-care therapy, or the participant declines standard-of-care therapy, or the participant did not tolerate standard-of-care therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* Evaluable disease (for participants in the Part 1 Dose Escalation) or measurable disease as per RECIST v1.1 (for participants in the Part 2 Dose Expansion).
* Acceptable organ function at Screening.
* Acceptable hematologic function at Screening.
* Adequate coagulation parameters at Screening.
* Female participants of childbearing potential must:

  1. Have a negative pregnancy test (serum) at Screening.
  2. Agree to use at least one highly effective form of contraception during study treatment and after the last dose of ORM-5029.
* Male participants with female partners of childbearing potential must:

  1. Agree to use at least one highly effective form of contraception during study treatment and after the last dose of ORM-5029.
  2. Refrain from donating sperm during their participation in the study and after the last dose of ORM-5029.
* Resolution of all toxicities of prior therapy or surgical procedures to baseline or Grade 1 (except for neuropathy, which must have resolved to Grade ≤2, hypothyroidism requiring medication, and alopecia).
* Adequate cardiac left ventricular function, as defined by a left ventricular ejection fraction (LVEF) ≥ institutional standard of normal.
* Life expectancy of ≥12 weeks according to the Investigator's judgment.

KEY EXCLUSION CRITERIA

* Systemic antineoplastic agent or radiation therapy given within 14 days prior to the first dose of ORM-5029.
* Known sensitivity to any of the ingredients of ORM-5029, including previously reported infusion reactions to pertuzumab leading to pertuzumab treatment discontinuation.
* History of other malignancy within the last 2 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome.
* Symptomatic central nervous system (CNS) metastases or presence of leptomeningeal disease. Participant with previously treated brain metastases may participate.
* Pregnant or breastfeeding.
* Major surgery (excluding placement of vascular access) within 4 weeks prior to first dose of ORM-5029.
* Uncontrolled hypertension (systolic BP ≥160 mmHg; diastolic BP ≥100 mmHg) despite adequate treatment prior to the first dose of ORM-5029.
* Cardiac diseases currently or within the last 6 months as defined by New York Heart Association ≥Class 2.
* Mean resting QT interval corrected for heart rate (QTc) interval using the Fridericia formula (QTcF) >450 msec for males and >470 msec for females.
* Concurrent treatment with medications that are well-known to prolong the QT interval (see CredibleMeds website: https://www.crediblemeds.org/) unless a participant is QT stable on QT prolonging medication for at least 4 weeks.
* Severe dyspnea at rest, due to complications of advanced malignancy.
* Past medical history or complications of interstitial lung disease. Note: Participants with history of radiation induced interstitial lung disease may be enrolled if the participant's symptoms have recovered
* Active, uncontrolled bacterial, fungal, or viral infection, including known hepatitis B virus (HBV), known hepatitis C virus (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.

  1. HIV Seropositive participants who are healthy and at low risk for AIDS-related outcomes can be considered eligible. HIV positive participants must be evaluated and discussed with the Medical Monitor, and should have:

     * CD4+ (cluster of differentiation 4) T-cell counts ≥350 cells/μL
     * No prior history of AIDS-defining opportunistic infections
     * Received established anti-retroviral therapy for at least four weeks and have an HIV viral load <400 copies/mL prior to enrolment.
  2. Participants who are hepatitis B surface antigen positive are eligible if they have received HBV antiviral therapy for at least 4 weeks prior to the first dose of ORM-5029 and have undetectable HBV viral load prior to enrolment. Note: Participants must remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.
  3. Participants with a history of HCV infection are eligible if they have received curative treatment and HCV viral load is undetectable prior to enrolment. Participants who are HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution are eligible. Note: Participants must have completed curative antiviral therapy at least 4 weeks prior to enrolment.
* Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease (with exception of participants with Gilbert's Syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per Investigator assessment).
* Moderate or severe hepatic impairment (i.e., Child-Pugh class B or C).
* Any bleeding disorder (e.g., coagulopathy) or history of chronic bleeding and participants on therapeutic anticoagulant therapy during the treatment. Note: Participants on prophylactic anticoagulant therapy are considered eligible.
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) and Expansion Dose Level (EDL) [Dose Escalation Only] | DLT assessment period: At the end of Cycle 1 (each cycle is 21 or 28 days); Approximately 18 months for MTD and EDL
  Identify the Dose-limiting Toxicities (DLTs) for each dose level tested and determine the MTD and EDL for ORM-5029
Incidence of Adverse Events (AEs) | Every cycle (each cycle is 21 or 28 days) until study discontinuation; Approximately 30 months
  Evaluate the safety and tolerability of ORM-5029 by identifying the treatment-emergent adverse events (TEAEs)
Define the Objective Response Rate (ORR) of ORM-5029 based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 [Dose Expansion Only] | Approximately 30 months
  ORR is defined as the percentage of subjects with Partial Response (PR) or Complete Response (CR)
Define the Duration of Response (DOR) of ORM-5029 based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 [Dose Expansion Only] | Approximately 30 months
  DOR is defined as the length of time from the date of the first documented response (PR or CR) until the date of first documented progression or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Assess pharmacokinetic (PK) parameters including area under the concentration versus time curve from time 0 hours to the last quantifiable concentration (AUC0-last) and from time 0 hours to infinity (AUC0-inf) | Serial PK collections at on Days 1, 2, 4, 8 and 15 of Cycle 1 and Day 1 of Cycle 3 (Pre-dose and at multiple timepoints [up to 6 hours]; each cycle is 21 or 28 days)
Assess maximum plasma and serum drug concentration (Cmax) | Serial PK collections at on Days 1, 2, 4, 8 and 15 of Cycle 1 and Day 1 of Cycle 3 (Pre-dose and at multiple timepoints [up to 6 hours]; each cycle is 21 or 28 days)
Define time to Cmax (Tmax) | Serial PK collections at on Days 1, 2, 4, 8 and 15 of Cycle 1 and Day 1 of Cycle 3 (Pre-dose and at multiple timepoints [up to 6 hours]; each cycle is 21 or 28 days)
Access pharmacokinetic (PK) parameters including terminal rate consent and terminal elimination half-life (t1/2) | Serial PK collections at Baseline, Days 2, 4, 8 and 15 of Cycle 1 and Day 1 of Cycle 3 (Pre-dose and at multiple timepoints [up to 6 hours]; each cycle is 21 or 28 days)
Define Clinical Benefit Rate (CBR) of ORM-5029 based on RECIST 1.1 | Approximately 30 months
  CBR is defined as CR + PR + stable disease (SD) up to 4 months
Define Time to Response (TTR) of ORM-5029 based on RECIST 1.1 | Approximately 30 months
  TTR is defined as the length of time from baseline until the date of first documented response (PR or CR)
Define Duration of Response (DOR) of ORM-5029 based on RECIST 1.1 [Dose Escalation Only] | Approximately 30 months
  DOR is defined as the length of time from the date of the first documented response (PR or CR) until the date of first documented progression or date of death from any cause, whichever came first
Assess Progression-free survival (PFS) of ORM-5029 based on RECIST 1.1 | Approximately 30 months
  PFS is defined as the length of time from baseline until the date of first documented progression or date of death from any cause, whichever came first
Assess overall survival (OS) | Following study discontinuation until withdrawal for any reason or death; Approximately 30 months
Incidence of anti-drug antibody (ADA) against ORM-5029 | Sample collection at Baseline, Day 1 of every Cycle until study discontinuation (each cycle is 21 or 28 days); Approximately 30 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine-New York, New York, New York
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology - Virginia Cancer Specialists, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No